CLINICAL TRIAL: NCT04463251
Title: International, Double Blind, Randomized, Placebo-controlled Study to Evaluate the Effect on Parameters of Systemic Inflammation and Disease Outcomes and Safety of RPH-104 in Subjects With Acute ST-elevation Myocardial Infarction
Brief Title: Study to Evaluate the Effect on Parameters of Systemic Inflammation and Disease Outcomes and Safety of RPH-104 in Subjects With Acute ST-elevation Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm Overseas, Inc. (Industry)
Collaborators: Cromos Pharma LLC (Industry); Data Management 365 (Industry); Keystat, LLC (Industry); R-Pharm (Industry); K-Research, LLC (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04018075
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
Keywords: STEMI; Myocardial infarction; Cardiovascular diseases; CVD; Coronary heart disease; CHD
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RPH-104 80 mg (Experimental): subjects received subcutaneous single injection of 2 mL (80 mg) of RPH-104 and 2 mL of placebo on different administration sites
  Interventions: Biological: RPH-104 80 mg; Drug: Placebo
- RPH-104 160 mg (Experimental): subjects received subcutaneous single injection of 2 mL (80 mg) of RPH-104 and 2 mL of (80 mg) of RPH-104 on different administration sites
  Interventions: Biological: RPH-104 80 mg
- Placebo (Placebo Comparator): subjects received subcutaneous single injection of 2 mL of placebo and 2 mL of placebo on different administration sites
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RPH-104 80 mg — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL transparent glass vial
  Other Names: goflikicept
  Arms: RPH-104 160 mg; RPH-104 80 mg
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution for Injection), 2 mL in the 4-mL transparent glass vial
  Arms: Placebo; RPH-104 80 mg

SUMMARY:
The goal of the study was to evaluate the effect of single administration of RPH-104 at 80 mg and 160 mg on parameters of systemic inflammation and outcomes of the disease in subjects with ST-segment elevation myocardial infarction (STEMI)

DETAILED DESCRIPTION:
After signing the informed consent form, the investigator assessed the subject's eligibility for the study. The following procedures were performed during the screening: collection of medical history, recording previous and concomitant therapy, demographic data, recording 12-lead ECG findings on which STEMI diagnosis was based, recording date and time of STEMI symptom development, recording date, time and results of coronary angiography (CAG) at admission to the study site, measurement of blood neutrophil count, vital signs, physical examination including measurement of body weight (if hospital bed is available), blood sampling for hematology, biochemistry, determination of concentration of hsCRP and brain natriuretic peptide (BNP; N-terminal (NT)-pro hormone brain natriuretic peptide (NT-pro-BNP)), for females with retained reproductive potential - pregnancy test (test strips).

The subjects meeting selection criteria were randomized to one of the three groups (in 1:1:1 ratio) for single subcutaneous administration of RPH-104 80 mg, RPH-104 160 mg or placebo.

Screening, randomization and administration of the study products were made on the same (first) study day.

Further 4-week (28-day) clinical follow-up and additional 6- and 12-month clinical follow-up period were performed.

The end of clinical part of the study was the date of the last visit of the last subject within additional 12-month clinical follow-up.

The maximum number of screened patients was planned to be 146 subjects, 102 subjects were randomized, 34 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who gave voluntary written Informed consent to participate in the study and to follow all Protocol procedures.
* STEMI diagnosis defined as chest pain or its equivalent with ECG findings evidencing ST elevation (>1 mm) in two or more consecutive leads or acute left bunch branch block according the investigator's judgement.
* Percutaneous coronary intervention (PCI) with stenting was performed within no more than 12 hours after onset of chest pain or its equivalent and randomization was performed in no more than 12 hours after PCI (overall within 24 hours of onset of chest pain or equivalent).
* Consent of female subjects with childbearing potential defined as all female subjects with physiological potential to conceive, to use highly effective contraceptive methods throughout the study starting from screening (signing Informed Consent Form) and negative pregnancy test.

Highly effective contraceptive methods include combination of two of the following methods (a+b or a+c or b+c):

1. oral, injection or implanted hormonal contraceptives; in case of oral contraceptives, the female subjects should administer the same product for at least 3 months prior to the study therapy;
2. intrauterine device or contraceptive system;
3. barrier methods: condom or occlusive cap (diaphragm or cervical cap / vaginal fornix cap) with spermicidal foam/gel/film/cream/vaginal suppository

   * Ability and willingness of the subject, according to the reasonable investigator's judgment, to attend the study site at all scheduled visits, undergo the study procedures and follow the Protocol requirements including subcutaneous injections by qualified site personnel.

Exclusion Criteria:

* Hypersensitivity to test product (RPH-104) and/or its ingredients/excipients.
* Pregnancy and breastfeeding.
* Verified chronic heart failure (The American Heart Association / The American College of Cardiology (AHA/ACC) C-D class, New York Heart Association (NYHA) Functional class (FC) III-IV)
* Pre-existing severe valvular heart disease according to the investigator's assessment.
* Pre-existing left ventricular (LV) dysfunction (ejection fraction (EF)<40%)
* History of STEMI
* Complications of acute myocardial infarction (MI) in the form of acute left ventricular failure and cardiogenic shock defined as stable blood pressure decrease (SBP<90 mm Hg) associated with signs of hypoperfusion as well as cases when inotropic and/or mechanical support is required to maintain SBP; and / or unstable hemodynamics.
* Active infections (acute or chronic); active tuberculosis.
* Recent (less than 5 half-life periods) or current administration of colchicine, as well as agents with an immunosuppressant mechanism of action, including, but not limited to:

glucocorticoids at doses of > 1 mg/kg of methylprednisolone equivalent, tumor necrosis factor-alfa (TNFα) blockers, Interleukin-1 (IL-1) and other biological drugs, cyclosporine and other immunosuppressants. Non-steroidal anti-inflammatory drugs (NSAIDs) are allowed.

* Immunization with live vaccines within 90 days prior to the study product administration.
* Chronic systemic autoimmune or autoinflammatory diseases
* Suspected necessity in cardiosurgery.
* Oncology (or diagnosis of oncology within the last 5 years).
* History of organ transplantation or necessity in transplantation at the screening initiation or scheduled transplantation during the study.
* Neutropenia (absolute neutrophil count <1800/mm^3).
* Participation in another clinical study within the previous 3 months prior to Screening visit.
* Other medical (including mental) conditions or abnormal laboratory findings which may increase the risk for the subject associated with the study participation or administration of the study products or which may affect interpretation of the study results and, according to the investigator, render the subject ineligible for the study.*

  *If, in the Investigator's opinion, administration of a non-live COVID-19 (SARS-CoV-2) vaccine increases the risk for the patient related to his/her participation in the study, the Investigator can make a decision not to include this patient into the study.
* The subjects working at the study site or subjects working for Sponsor directly involved in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lavrovsky, Study Director — R-Pharm Overseas, Inc.
Locations (11):
- United States (3):
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia Health System, Charlottesville, Virginia
  - VCU Health-Virginia Commonwealth University Health, Richmond, Virginia
- Russia (8):
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital named after V.V. Vinogradov of Moscow Healthcare Department", Moscow
  - State Institution of Healthcare in Moscow "City Clinical Hospital № 51 Moscow Health Department", Moscow
  - Federal State Budgetary Institution "National Medical Research Center for Cardiology" of the Ministry of Healthcare of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital named after V.V. Veresaev of Moscow Healthcare Department", Moscow
  - State Autonomous Healthcare Institution of the Perm Territory "City Clinical Hospital No. 4", Perm
  - Ryazan State Medical University n.a. academician I.P. Pavlov on the basis of Regional Clinical cardiology Dispensary, Ryazan
  - St. Petersburg State Budgetary Healthcare Institution "Saint Martyr Elizabeth City Hospital", Saint Petersburg
  - The State Budgetary Health Care Institution of the Yaroslavl Region "Regional Clinical Hospital", Yaroslavl

REFERENCES:
- [Derived] Abbate A, Van Tassell B, Bogin V, Markley R, Pevzner DV, Cremer PC, Meray I, Privalov DV, Taylor A, Grishin SA, Egorova AN, Ponomar EG, Lavrovsky Y, Samsonov MY; RPH-104 STEMI Study Investigators. Results of International, Double-Blind, Randomized, Placebo-Controlled, Phase IIa Study of Interleukin-1 Blockade With RPH-104 (Goflikicept) in Patients With ST-Segment-Elevation Myocardial Infarction (STEMI). Circulation. 2024 Aug 13;150(7):580-582. doi: 10.1161/CIRCULATIONAHA.124.069396. Epub 2024 Aug 12. No abstract available. PMID 39133774
- [Derived] Samsonov M, Bogin V, Van Tassell BW, Abbate A. Interleukin-1 blockade with RPH-104 in patients with acute ST-elevation myocardial infarction: study design and rationale. J Transl Med. 2021 Apr 26;19(1):169. doi: 10.1186/s12967-021-02828-z. PMID 33902621

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 11 sites (Russia - 8, USA - 3). A total of 102 patients were randomized. The safety set included all randomized patients.The full analysis set for efficacy analysis (FAS) included 101 patients (who received the study products and underwent at least one hsCRP measurement after administration of the study products. The Per Protocol Set (PPS) included 92 subjects from the FAS without significant protocol deviations affecting assessment of the primary efficacy parameter.
Period: Overall Study
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Started | 34 | 34 | 34
Safety Set | 34 | 34 | 34
Full Analysis Set (One patient in the Placebo arm was excluded from FAS population due to absence of High-sensitivity C-reactive protein (hsCRP) baseline measurement (the central laboratory was notable to perform an assay due to hemolysis)) | 34 | 34 | 33
Per Protocol Set | 30 | 31 | 31
Completed the Study Per Protocol | 33 | 30 | 31
Completed | 33 | 30 | 31
Not Completed | 1 | 4 | 3
Not completed — Death | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 33 | 101
Age, Continuous [Mean (Full Range); unit: years] | 58.9 [33 to 79] | 58.7 [38 to 86] | 59.3 [23 to 88] | 59 [23 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 12 | 28
  Male | 23 | 29 | 21 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 0 | 1
  Race: Black or African American | 3 | 0 | 0 | 3
  Race: White | 29 | 34 | 33 | 96
  Race: Hispanic | 1 | 0 | 0 | 1
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 28.7 [20.7 to 39.2] | 29.4 [20.3 to 49.1] | 30.3 [22.3 to 42.0] | 29.5 [20.3 to 49.1]

OUTCOME MEASURES:

1. Primary Outcome: High-sensitive С-reactive Protein (hsCRP) Area Under Curve (AUC) From Baseline Until Day 14 (Multiple Imputation Procedure)
Description: hsCRP area under curve (AUC) from baseline (Day 1) until Day 14
Time Frame: Day 1 until Day 14
Population: Full analysis set for efficacy analysis included all randomized subjects who received the study products (RPH-104 or placebo), and underwent at least one hsCRP measurement after administration of the study products. The FAS was the main population for efficacy assessment.
  Multiple imputation procedure was performed for hsCRP values which were missed on Day 14.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Groups:
- RPH-104 80 mg: subjects receive subcutaneous single injection of 2 mL (80 mg) of RPH-104 and 2 mL of placebo on different administration sites
  RPH-104 80 mg: solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL transparent glass vial
  Placebo: Normal Saline (0.9% Sodium Chloride solution for Injection), 2 mL in the 4-mL transparent glass vial
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
mg*day/L | 106.84 [79.72 to 143.19] | 107.65 [80.10 to 144.68] | 184.30 [136.06 to 249.65]
Statistical Analysis 1: Comparison: RPH-104 80 mg vs Placebo; The following (two-sided) hypotheses were tested: * Null hypothesis H0: the ratio of the geometric mean of hsCRP-AUC(days 1-14) in RPH-104 group to the geometric mean of hsCRP-AUC(days 1-14) in the placebo group is equal to 1. * Alternative hypothesis H1: the ratio of the geometric mean of hsCRP-AUC(days 1-14) in RPH-104 group to the geometric mean of hsCRP-AUC(days 1-14) in the placebo group is different from 1; Test type: Other; Least square means ratio = 0.58, 95% CI 2-sided [0.37 to 0.91] — Least square means ratio with two-sided Dunnett's adjusted 95% CI for RPH-104 80 mg / Placebo. Ratio was calculated instead of difference because log data transformation
Statistical Analysis 2: Comparison: RPH-104 160 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.58, 95% CI 2-sided [0.37 to 0.91] — Least square means ratio with two-sided Dunnett's adjusted 95% CI for RPH-104 160 mg / Placebo. Ratio was calculated instead of difference because log data transformation

2. Primary Outcome: High-sensitive С-reactive Protein (hsCRP) Area Under Curve (AUC) From Baseline Until Day 14 (сomplete Cases)
Description: hsCRP area under curve (AUC) from baseline (Day 1) until Day 14
Time Frame: Day 1 until Day 14
Population: Full analysis set for efficacy analysis included all randomized subjects who received the study products (RPH-104 or placebo), and underwent at least one hsCRP measurement after administration of the study products. The FAS was the main population for efficacy assessment.
  The model included patients with complete data (complete cases) in the FAS population. No data imputations were performed.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
mg*day/L | 96.72 [70.57 to 132.54] | 106.71 [77.53 to 146.87] | 178.59 [129.54 to 246.21]
Statistical Analysis 1: Comparison: RPH-104 80 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.54, 95% CI 2-sided [0.34 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RPH-104 160 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.60, 95% CI 2-sided [0.37 to 0.95] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: High-sensitive С-reactive Protein (hsCRP) Area Under Curve (AUC) From Baseline Until Day 14 (Sensitivity Analysis, Multiple Imputation Procedure)
Description: hsCRP area under curve (AUC) from baseline (Day 1) until Day 14 (sensitivity analysis)
Time Frame: Day 1 until Day 14
Population: At the stage of final analysis, sensitivity analysis was performed for the per protocol population (PPS).
  Multiple imputation procedure was performed for hsCRP values which were missed on Day 14.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 30 | 31 | 31
mg*day/L | 96.57 [69.75 to 133.71] | 105.30 [76.00 to 145.91] | 173.48 [124.31 to 242.10]
Statistical Analysis 1: Comparison: RPH-104 80 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.56, 95% CI 2-sided [0.34 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RPH-104 160 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.61, 95% CI 2-sided [0.38 to 0.98] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: High-sensitive С-reactive Protein (hsCRP) Area Under Curve (AUC) From Baseline Until Day 14 (Sensitivity Analysis, Complete Cases)
Description: hsCRP area under curve (AUC) from baseline (Day 1) until Day 14 (sensitivity analysis)
Time Frame: Day 1 until Day 14
Population: At the stage of final analysis, sensitivity analysis was performed for the per protocol population (PPS).
  The model included patients with complete data (complete cases) in the PPS population. No data imputations were performed.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 30 | 31 | 31
mg*day/L | 95.35 [68.41 to 132.91] | 104.26 [75.07 to 144.81] | 171.69 [122.74 to 240.16]
Statistical Analysis 1: Comparison: RPH-104 80 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.56, 95% CI 2-sided [0.34 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RPH-104 160 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least square means ratio = 0.61, 95% CI 2-sided [0.38 to 0.98] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: hsCRP AUC From Baseline Until Day 28 (Multiple Imputation Procedure)
Description: hsCRP AUC from baseline (Day 1) until Day 28
Time Frame: up to Day 28
Population: Full analysis set for efficacy analysis included all randomized subjects who received the study products (RPH-104 or placebo), and underwent at least one hsCRP measurement after administration of the study products. The FAS was the main population for efficacy assessment.
  Multiple imputation procedure was performed for hsCRP values which were missed on Day 28.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
mg*day/L | 148.58 [111.62 to 197.79] | 136.84 [102.44 to 182.78] | 285.78 [212.21 to 384.86]
Statistical Analysis 1: Comparison: RPH-104 80 mg vs Placebo; The following (two-sided) hypotheses were tested: Null hypothesis H0: the ratio of the geometric mean of hsCRP-AUC(days 1-28) in RPH-104 group to the geometric mean of hsCRP-AUC(days 1-28) in the placebo group is equal to 1. Alternative hypothesis H1: the ratio of the geometric mean of hsCRP-AUC(days 1-28) in RPH-104 group to the geometric mean of hsCRP-AUC(days 1-28) in the placebo group is different from 1; Test type: Other; Least square means ratio = 0.52, 95% CI 2-sided [0.34 to 0.81]; Least square means ratio with two-sided Dunnett's adjusted 95% CI for RPH-104 80 mg / Placebo. Ratio was calculated instead of difference because log data transformation
Statistical Analysis 2: Comparison: RPH-104 160 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other; Least square means ratio = 0.48, 95% CI 2-sided [0.31 to 0.74] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: hsCRP AUC From Baseline Until Day 28 (Complete Cases)
Description: hsCRP AUC from baseline (Day 1) until Day 28
Time Frame: up to Day 28
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
mg*day/L | 130.07 [95.41 to 177.31] | 131.27 [95.95 to 179.60] | 277.13 [202.68 to 378.94]
Statistical Analysis 1: Comparison: RPH-104 80 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other; Least square means ratio = 0.47, 95% CI 2-sided [0.29 to 0.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RPH-104 160 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Other; Least square means ratio = 0.47, 95% CI 2-sided [0.30 to 0.75] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Number of Patients With Fatal Outcomes (Cardiac and Non-cardiac) During 12-month Follow-up Period
Description: Any fatal outcomes were evaluated by the investigators and Independent study outcome assessment committee (ISOAC). ISOAC assessments were considered as the main data for conclusions, the investigator's assessments were presented for informational purposes only.
Time Frame: up to Day 365
Population: Analysis was performed at the stage of final analysis for the FAS population. Data for fatal cases (deaths) were derived from CRF records. The CRF provided "Yes", "No" and "Unknown" for patient's alive status. Unknown was naturally missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
Participants
  Cardiovascular death | 1 | 0 | 1
  Non-cardiovascular death | 0 | 0 | 0
  Patient is alive | 33 | 31 | 30
  Unknown | 0 | 3 | 2

8. Secondary Outcome: Number of Patients With of Hospitalizations Due to Heart Failure (HF) or Other Cardiac Reasons Not Associated With HF, or Due to Non-cardiac Reasons During 12-month Follow-up Period
Description: Number of patients with hospitalizations for any reason during 12-month follow-up period, assessed by ISOAC.
Time Frame: up to Day 365
Population: Analysis was performed at the stage of final analysis for the FAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
Participants
  Hospitalization for cardiovascular reasons (except Heart Failure) | 2 | 0 | 3
  Hospitalization for new HF onset | 0 | 0 | 0
  Hospitalization due to non-cardiac reasons | 2 | 1 | 1
  Unknown (premature discontinuation) | 0 | 3 | 2

9. Secondary Outcome: Number of Patients With New Cases of HF During 12-month Follow-up Period
Description: New cases of HF are defined as hospitalization due to HF or an emergency outpatient visit due to heart failure.
  ISOAC assessment
Time Frame: up to Day 365
Population: FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
Participants | 0 | 0 | 0

10. Secondary Outcome: Changes in Levels of Brain Natriuretic Peptide (BNP) During 12-month Follow-up Period Compared to Baseline
Description: Change in levels of BNP during 12-month follow-up period compared to baseline. (Brain Natriuretic Peptide (BNP) was measured in pmol/L.) Increased levels of BNP can be considered as marker of hemodynamic stress and surrogate marker of Heart Failure.
  The reported Least square means and confidence interval were from a repeated measures model on log transformed BNP data containing treatment, visit as factors, log baseline BNP as a continuous covariate and treatment by visit as interaction terms. Due to log-transformed data, change from baseline was defined as division value at corresponding time point and baseline value, thus the smallest value of the change from baseline indicates a better outcome or improvement.
Time Frame: From Day 1 until Day 365
Population: Analysis was performed at the stage of final analysis for the FAS population. No data imputations were performed.
  Here, "Number Analyzed" indicates patients with assessable date each corresponding time point. Change from baseline was calculated for patients who had data at baseline and corresponding time point.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ratio
  Change from baseline (Day 3) | 1.74 [1.25 to 2.42] | 1.23 [0.88 to 1.71] | 1.62 [1.16 to 2.27]
  Change from baseline (Day 14): number analyzed (Participants) | 31 | 29 | 32
  Change from baseline (Day 14) | 2.04 [1.34 to 3.11] | 1.27 [0.83 to 1.94] | 1.52 [1.00 to 2.32]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 31 | 32 | 31
  Change from baseline (Day 28 / Early withdrawal) | 1.50 [1.50 to 2.37] | 1.05 [0.67 to 1.66] | 1.14 [0.72 to 1.81]
  Change from baseline (Month 12): number analyzed (Participants) | 33 | 27 | 29
  Change from baseline (Month 12) | 0.64 [0.40 to 1.05] | 0.44 [0.26 to 0.73] | 0.67 [0.40 to 1.10]

11. Secondary Outcome: Changes in End-diastolic (EDV) Volume After 12 Months Compared to Baseline
Description: Apical 4-, 2-, and 3-chamber view in B-mode: End-diastolic (EDV) volumes. Measured by echocardiography (Echo-CG) (in mL). The reported Least square means and confidence interval were from a repeated measures model on EDV data containing treatment, visit as factors, baseline EDV as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: FAS population. No data imputations were performed. Here, "Number Analyzed" indicates patients with assessable date each corresponding time point. Change from baseline was calculated for patients who had data at baseline and corresponding time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: ml
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ml
  Day 1 (Baseline): number analyzed (Participants) | 33 | 33 | 30
  Day 1 (Baseline) | 123.92 [115.80 to 132.04] | 123.10 [114.57 to 131.62] | 122.64 [114.11 to 131.18]
  Day 28 / Early withdrawal: number analyzed (Participants) | 31 | 29 | 31
  Day 28 / Early withdrawal | 123.32 [114.91 to 131.72] | 126.49 [117.52 to 135.47] | 132.34 [123.67 to 141.01]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 30 | 29 | 29
  Change from baseline (Day 28 / Early withdrawal) | -0.60 [-11.29 to 10.08] | 3.40 [-7.45 to 14.25] | 9.70 [-1.33 to 20.72]
  Month 12: number analyzed (Participants) | 32 | 28 | 29
  Month 12 | 112.80 [104.56 to 121.04] | 116.88 [107.77 to 125.99] | 119.98 [111.03 to 128.93]
  Change from baseline (Month 12): number analyzed (Participants) | 32 | 28 | 27
  Change from baseline (Month 12) | -11.12 [-22.86 to 0.62] | -6.22 [-18.41 to 5.97] | -2.66 [-15.20 to 9.88]

12. Secondary Outcome: BNP AUC From Day 1 (Baseline) Until Day 28
Time Frame: up to Day 28
Population: Full analysis set for efficacy analysis included all randomized subjects who received the study products (RPH-104 or placebo), and underwent at least one hsCRP measurement after administration of the study products. The FAS was the main population for efficacy assessment.
  The model included patients with complete data (complete cases).
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pmol*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
pmol*day/L | 923.04 [702.30 to 1213.18] | 833.55 [628.07 to 1106.27] | 954.22 [725.29 to 1255.42]

13. Secondary Outcome: NT-pro-BNP AUC From Day 1 (Baseline) Until Day 28
Time Frame: up to Day 28
Population: as for outcome 12
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pmol*day/L
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
pmol*day/L | 2152.07 [1591.94 to 2909.29] | 1940.71 [1438.84 to 2617.62] | 2597.13 [1928.48 to 3497.62]

14. Secondary Outcome: Number of Patients With Fatal Outcomes (Due to Any Reason) or Hospitalizations Due to HF or Emergency Outpatient Visits Due to HF During 12-month Follow-up Period
Description: ISOAC assessment
Time Frame: up to Day 365
Population: FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
Participants | 1 | 0 | 1

15. Secondary Outcome: Number of Patients With Fatal Outcomes (Due to Any Reason) or Hospitalizations Due to HF During 12-month Follow-up Period
Description: ISOAC assessment
Time Frame: up to Day 365
Population: FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
Participants | 1 | 0 | 1

16. Secondary Outcome: Changes in Levels of Brain Natriuretic Peptide (NT-proBNP) During 12-month Follow-up Period Compared to Baseline
Description: Change in levels of NT-proBNP during 12-month follow-up period compared to baseline.
  The reported Least square means and confidence interval were from a repeated measures model on log transformed NT-proBNP data containing treatment, visit as factors, log transformed baseline NT-proBNP as a continuous covariate and treatment by visit as interaction terms.
  For log-transformed data change was defined as division value at corresponding time point and baseline value.
Time Frame: From Day 1 until Day 365
Population: as for outcome 10
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ratio
  Change from baseline (Day 3): number analyzed (Participants) | 33 | 33 | 33
  Change from baseline (Day 3) | 2.24 [1.60 to 3.14] | 1.85 [1.32 to 2.58] | 2.32 [1.66 to 3.25]
  Change from baseline (Day 14): number analyzed (Participants) | 30 | 31 | 32
  Change from baseline (Day 14) | 1.70 [1.10 to 2.63] | 1.28 [0.83 to 1.96] | 1.59 [1.04 to 2.44]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 30 | 32 | 32
  Change from baseline (Day 28 / Early withdrawal) | 1.46 [0.90 to 2.37] | 1.28 [0.80 to 2.06] | 1.45 [0.90 to 2.34]
  Change from baseline (Month 12): number analyzed (Participants) | 32 | 28 | 29
  Change from baseline (Month 12) | 0.38 [0.23 to 0.64] | 0.37 [0.22 to 0.63] | 0.46 [0.27 to 0.78]

17. Secondary Outcome: Changes in End-systolic (ESV) Volume After 12 Months Compared to Baseline
Description: Apical 4-, 2-, and 3-chamber view in B-mode: End-systolic (ESV) volumes. Measured by echocardiography (Echo-CG) (in mL). The reported Least square means and confidence interval were from a repeated measures model on ESV data containing treatment, visit as factors, baseline ESV as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: ml
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ml
  Day 1 (Baseline): number analyzed (Participants) | 33 | 33 | 30
  Day 1 (Baseline) | 54.20 [48.76 to 59.65] | 54.60 [48.90 to 60.30] | 54.55 [48.86 to 60.24]
  Day 28 / Early withdrawal: number analyzed (Participants) | 31 | 29 | 31
  Day 28 / Early withdrawal | 52.30 [46.67 to 57.93] | 54.31 [48.32 to 60.30] | 52.07 [46.29 to 57.85]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 30 | 29 | 29
  Change from baseline (Day 28 / Early withdrawal) | -1.90 [-8.90 to 5.09] | -0.30 [-7.40 to 6.81] | -2.47 [-9.69 to 4.74]
  Month 12: number analyzed (Participants) | 32 | 28 | 29
  Month 12 | 45.88 [40.35 to 51.40] | 48.67 [42.58 to 54.75] | 48.67 [42.71 to 54.63]
  Change from baseline (Month 12): number analyzed (Participants) | 32 | 28 | 27
  Change from baseline (Month 12) | -8.33 [-16.06 to -0.59] | -5.94 [-13.97 to 2.10] | -5.88 [-14.15 to 2.39]

18. Secondary Outcome: Changes in Ejection Fraction (EF) After 12 Months Compared to Baseline
Description: Apical 4-, 2-, and 3-chamber view in B-mode: Ejection fraction (EF) (Simpson method).
  Measured by echocardiography (Echo-CG) (in percentage). The reported Least square means and confidence interval were from a repeated measures model on EF data containing treatment, visit as factors, baseline EF as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of blood
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
percentage of blood
  Day 1 (Baseline): number analyzed (Participants) | 33 | 33 | 30
  Day 1 (Baseline) | 56.93 [54.61 to 59.25] | 56.51 [54.12 to 58.89] | 56.62 [54.19 to 59.05]
  Day 28 / Early withdrawal: number analyzed (Participants) | 31 | 29 | 31
  Day 28 / Early withdrawal | 58.98 [56.57 to 61.39] | 58.35 [55.82 to 60.88] | 61.26 [58.79 to 63.73]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 30 | 29 | 29
  Change from baseline (Day 28 / Early withdrawal) | 2.05 [-2.02 to 6.13] | 1.84 [-2.27 to 5.96] | 4.64 [0.41 to 8.87]
  Month 12: number analyzed (Participants) | 32 | 28 | 29
  Month 12 | 60.87 [58.52 to 63.22] | 60.31 [57.74 to 62.88] | 61.17 [58.61 to 63.72]
  Change from baseline (Month 12): number analyzed (Participants) | 32 | 28 | 27
  Change from baseline (Month 12) | 3.94 [0.16 to 7.72] | 3.80 [-0.10 to 7.70] | 4.55 [0.52 to 8.58]

19. Secondary Outcome: Changes in Regional LV Function After 12 Months Compared to Baseline
Description: Apical 4-, 2-, and 3-chamber view in B-mode: assessment of regional LV function using the wall motion score index (WMSI), measured by Echo-CG.
  The wall motion score index was calculated by assigning each segment a score based on its systolic function (normal = 1 (the best), hypokinesis = 2, akinesis = 3, dyskinesis = 4 (the worst)). The WMSI is the sum of all segmental scores divided by the number of segments analyzed (scale 1 - 4). A wall motion score index of 1 is normal (the best outcome). The higher the wall motion score index the worse is the outcome.
  The reported Least square means and confidence interval were from a repeated measures model on Regional LV Function data containing treatment, visit as factors, baseline Regional LV Function data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: index units
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
index units
  Day 1 (Baseline): number analyzed (Participants) | 31 | 33 | 28
  Day 1 (Baseline) | 1.40 [1.32 to 1.48] | 1.39 [1.31 to 1.47] | 1.40 [1.32 to 1.49]
  Day 28 / Early withdrawal: number analyzed (Participants) | 25 | 28 | 29
  Day 28 / Early withdrawal | 1.23 [1.14 to 1.31] | 1.29 [1.20 to 1.37] | 1.21 [1.12 to 1.30]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 25 | 27 | 25
  Change from baseline (Day 28 / Early withdrawal) | -0.17 [-0.29 to -0.06] | -0.10 [-0.21 to 0.01] | -0.19 [-0.31 to -0.07]
  Month 12: number analyzed (Participants) | 21 | 16 | 14
  Month 12 | 1.19 [1.09 to 1.28] | 1.26 [1.15 to 1.37] | 1.17 [1.06 to 1.29]
  Change from baseline (Month 12): number analyzed (Participants) | 20 | 16 | 13
  Change from baseline (Month 12) | -0.21 [-0.34 to -0.08] | -0.13 [-0.27 to 0.01] | -0.23 [-0.38 to -0.08]

20. Secondary Outcome: Changes in Stroke Volume (SV) Compared to Baseline
Description: Apical 4-, 2-, and 3-chamber view in B-mode: assessment of Stroke Volume (SV), measured by Echo-CG.
  The reported Least square means and confidence interval were from a repeated measures model on SV data containing treatment, visit as factors, baseline SV data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: ml
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ml
  Day 1 (Baseline): number analyzed (Participants) | 33 | 33 | 30
  Day 1 (Baseline) | 70.09 [65.34 to 74.83] | 68.15 [63.22 to 73.07] | 67.61 [62.64 to 72.59]
  Day 28 / Early withdrawal: number analyzed (Participants) | 31 | 29 | 31
  Day 28 / Early withdrawal | 71.05 [66.11 to 75.99] | 71.62 [66.39 to 76.86] | 79.79 [74.72 to 84.86]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 30 | 29 | 29
  Change from baseline (Day 28 / Early withdrawal) | 0.96 [-6.18 to 8.10] | 3.48 [-3.75 to 10.71] | 12.17 [4.81 to 19.54]
  Month 12: number analyzed (Participants) | 32 | 28 | 29
  Month 12 | 66.09 [61.28 to 70.90] | 67.61 [62.31 to 72.91] | 70.63 [65.37 to 75.89]
  Change from baseline (Month 12): number analyzed (Participants) | 32 | 28 | 27
  Change from baseline (Month 12) | -4.00 [-11.38 to 3.38] | -0.54 [-8.19 to 7.11] | 3.02 [-4.88 to 10.91]

21. Secondary Outcome: Changes in Global Longitudinal Strain (GLS) Compared to Baseline
Description: Apical 4-, 2-, and 3-chamber view in B-mode: assessment of Global Longitudinal Strain (GLS), measured by Echo-CG.
  GLS is a measure of longitudinal shortening of the myocardium as a percentage (change in length as a proportion to baseline length), thus explaining the negative values.
  The reported Least square means and confidence interval were from a repeated measures model on GLS data containing treatment, visit as factors, baseline GLS data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of myocardial shortening
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
percentage of myocardial shortening
  Day 1 (Baseline): number analyzed (Participants) | 31 | 30 | 26
  Day 1 (Baseline) | -15.39 [-16.50 to -14.28] | -15.24 [-16.42 to -14.07] | -14.60 [-15.80 to -13.40]
  Day 28 / Early withdrawal: number analyzed (Participants) | 29 | 26 | 27
  Day 28 / Early withdrawal | -16.69 [-17.88 to -15.50] | -16.20 [-17.46 to -14.94] | -18.22 [-19.47 to -16.96]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 27 | 26 | 24
  Change from baseline (Day 28 / Early withdrawal) | -1.30 [-3.03 to 0.43] | -0.96 [-2.72 to 0.81] | -3.62 [-5.48 to -1.76]
  Month 12: number analyzed (Participants) | 28 | 21 | 24
  Month 12 | -17.80 [-18.99 to -16.62] | -18.16 [-19.54 to -16.78] | -19.47 [-20.81 to -18.13]
  Change from baseline (Month 12): number analyzed (Participants) | 27 | 21 | 21
  Change from baseline (Month 12) | -2.41 [-4.20 to -0.63] | -2.91 [-4.85 to -0.98] | -4.87 [-6.86 to -2.87]

22. Secondary Outcome: Changes of Fractional Area Change (FAC) Compared to Baseline
Description: Right atrium and ventricle assessment from the apical 4-chamber right ventricular-focused view (with maximal right ventricular basal dimension) in B-mode and M-mode: Fractional Area Change (FAC).
  The reported Least square means and confidence interval were from a repeated measures model on FAC data containing treatment, visit as factors, baseline FAC data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of area
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
percentage of area
  Day 1 (Baseline): number analyzed (Participants) | 20 | 27 | 19
  Day 1 (Baseline) | 48.65 [45.11 to 52.19] | 48.45 [45.25 to 51.65] | 48.93 [45.30 to 52.56]
  Day 28 / Early withdrawal: number analyzed (Participants) | 20 | 20 | 20
  Day 28 / Early withdrawal | 51.73 [47.73 to 55.74] | 50.78 [47.03 to 54.53] | 50.27 [46.34 to 54.19]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 16 | 19 | 16
  Change from baseline (Day 28 / Early withdrawal) | 3.09 [-2.78 to 8.95] | 2.33 [-2.90 to 7.56] | 1.34 [-4.59 to 7.26]
  Month 12: number analyzed (Participants) | 22 | 18 | 16
  Month 12 | 49.22 [44.45 to 53.98] | 51.32 [46.97 to 55.66] | 48.15 [43.13 to 53.16]
  Change from baseline (Month 12): number analyzed (Participants) | 11 | 14 | 10
  Change from baseline (Month 12) | 0.57 [-6.07 to 7.21] | 2.87 [-2.98 to 8.72] | -0.78 [-7.75 to 6.18]

23. Secondary Outcome: Changes in Tricuspid Annular Plane Systolic Excursion (TAPSE) Parameter Compared to Baseline
Description: Right atrium and ventricle assessment from the apical 4-chamber right ventricular-focused view (with maximal right ventricular basal dimension) in B-mode and M-mode: tricuspid annular plane systolic excursion (TAPSE).
  The reported Least square means and confidence interval were from a repeated measures model on TAPSE data containing treatment, visit as factors, baseline TAPSE data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Groups:
- Placebo: subjects received subjects received subcutaneous single injection of 2 mL of placebo and 2 mL of placebo on different administration sites
  Placebo: Normal Saline (0.9% Sodium Chloride solution for Injection), 2 mL in the 4-mL transparent glass vial
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
mm
  Day 1 (Baseline): number analyzed (Participants) | 24 | 29 | 28
  Day 1 (Baseline) | 21.87 [20.46 to 23.29] | 21.76 [20.43 to 23.08] | 21.19 [19.87 to 22.51]
  Day 28 / Early withdrawal: number analyzed (Participants) | 28 | 28 | 28
  Day 28 / Early withdrawal | 22.09 [20.61 to 23.56] | 22.71 [21.22 to 24.21] | 22.79 [21.37 to 24.21]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 22 | 23 | 24
  Change from baseline (Day 28 / Early withdrawal) | 0.21 [-2.08 to 2.50] | 0.96 [-1.22 to 3.13] | 1.60 [-0.57 to 3.76]
  Month 12: number analyzed (Participants) | 27 | 20 | 27
  Month 12 | 21.88 [20.40 to 23.36] | 21.05 [19.42 to 22.69] | 22.71 [21.26 to 24.16]
  Change from baseline (Month 12): number analyzed (Participants) | 22 | 19 | 23
  Change from baseline (Month 12) | 0.00 [-2.29 to 2.30] | -0.70 [-3.01 to 1.60] | 1.52 [-0.68 to 3.72]

24. Secondary Outcome: Changes in Early Diastolic Transmitral Flow Velocity (E Velocity) Compared to Baseline
Description: Assessment of diastolic and systolic function, apical 4-chamber view in pulse-wave Doppler mode, tissue Doppler mode: Transmitral flow, pulsed wave (PW) Doppler, E.
  The reported Least square means and confidence interval were from a repeated measures model on E velocity data containing treatment, visit as factors, baseline E velocity data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
m/s
  Day 1 (Baseline): number analyzed (Participants) | 33 | 32 | 30
  Day 1 (Baseline) | 0.72 [0.67 to 0.77] | 0.70 [0.65 to 0.75] | 0.70 [0.65 to 0.75]
  Day 28 / Early withdrawal: number analyzed (Participants) | 32 | 30 | 31
  Day 28 / Early withdrawal | 0.72 [0.67 to 0.77] | 0.69 [0.63 to 0.74] | 0.79 [0.74 to 0.84]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 31 | 28 | 29
  Change from baseline (Day 28 / Early withdrawal) | -0.00 [-0.09 to 0.08] | -0.01 [-0.10 to 0.08] | 0.09 [-0.00 to 0.18]
  Month 12: number analyzed (Participants) | 32 | 27 | 30
  Month 12 | 0.67 [0.62 to 0.72] | 0.70 [0.64 to 0.75] | 0.76 [0.71 to 0.82]
  Change from baseline (Month 12): number analyzed (Participants) | 31 | 26 | 27
  Change from baseline (Month 12) | -0.05 [-0.13 to 0.03] | -0.00 [-0.09 to 0.08] | 0.06 [-0.02 to 0.14]

25. Secondary Outcome: Changes in Mitral Valve (MV) e'Sept Compared to Baseline
Description: Assessment of diastolic and systolic function, apical 4-chamber view in pulse-wave Doppler mode, tissue Doppler mode: Tissue Doppler Imaging, MV e'sept. Unit of measure is centimeter/second (cm/s). This is one of the diastolic function parameters (septal velocity fibrous ring of the mitral valve (MV)).
  The reported Least square means and confidence interval were from a repeated measures model on MV e'Sept data containing treatment, visit as factors, baseline MV e'Sept data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/s
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
cm/s
  Day 1 (Baseline): number analyzed (Participants) | 32 | 32 | 29
  Day 1 (Baseline) | 7.17 [6.68 to 7.67] | 7.14 [6.62 to 7.65] | 6.69 [6.17 to 7.21]
  Day 28 / Early withdrawal: number analyzed (Participants) | 31 | 31 | 30
  Day 28 / Early withdrawal | 6.47 [5.96 to 6.99] | 7.03 [6.49 to 7.57] | 7.09 [6.55 to 7.63]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 29 | 29 | 27
  Change from baseline (Day 28 / Early withdrawal) | -0.70 [-1.46 to 0.06] | -0.11 [-0.87 to 0.65] | 0.40 [-0.39 to 1.18]
  Month 12: number analyzed (Participants) | 30 | 28 | 29
  Month 12 | 6.51 [5.98 to 7.04] | 7.11 [6.55 to 7.68] | 7.11 [6.55 to 7.67]
  Change from baseline (Month 12): number analyzed (Participants) | 28 | 26 | 25
  Change from baseline (Month 12) | -0.66 [-1.45 to 0.13] | -0.02 [-0.83 to 0.79] | 0.42 [-0.42 to 1.26]

26. Secondary Outcome: Changes in Mitral Valve e'Lat Compared to Baseline
Description: Assessment of diastolic and systolic function, apical 4-chamber view in pulse-wave Doppler mode, tissue Doppler mode: Tissue Doppler Imaging, MV e'lat. Unit of measure is centimeter/second (cm/s). This is one of the diastolic function parameters (lateral velocity of fibrous ring of the mitral valve (MV)).
  The reported Least square means and confidence interval were from a repeated measures model on MV e'Lat data containing treatment, visit as factors, baseline MV e'Lat data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/s
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
cm/s
  Day 1 (Baseline): number analyzed (Participants) | 32 | 30 | 29
  Day 1 (Baseline) | 9.04 [8.32 to 9.76] | 9.04 [8.28 to 9.81] | 8.76 [8.01 to 9.51]
  Day 28 / Early withdrawal: number analyzed (Participants) | 30 | 31 | 29
  Day 28 / Early withdrawal | 9.55 [8.79 to 10.31] | 8.86 [8.06 to 9.67] | 9.61 [8.81 to 10.40]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 28 | 27 | 26
  Change from baseline (Day 28 / Early withdrawal) | 0.51 [-0.61 to 1.64] | -0.18 [-1.33 to 0.97] | 0.85 [-0.32 to 2.02]
  Month 12: number analyzed (Participants) | 31 | 28 | 29
  Month 12 | 9.24 [8.49 to 9.99] | 9.83 [9.00 to 10.66] | 9.63 [8.82 to 10.44]
  Change from baseline (Month 12): number analyzed (Participants) | 29 | 25 | 25
  Change from baseline (Month 12) | 0.20 [-0.94 to 1.35] | 0.79 [-0.42 to 2.00] | 0.87 [-0.35 to 2.09]

27. Secondary Outcome: Changes in Left Ventricular Stroke Volume (LV SV) Compared to Baseline
Description: Assessment of diastolic and systolic function, apical 4-chamber view in pulse-wave Doppler mode, tissue Doppler mode: LV outflow tract velocity-time integral (VTI) + Diameter. Tissue Doppler Imaging, LV Stroke Volume (pulse-wave Doppler mode).
  The reported Least square means and confidence interval were from a repeated measures model on LV SV data containing treatment, visit as factors, baseline LV SV data as a continuous covariate and treatment by visit as interaction terms.
Time Frame: From Day 1 Until Day 365
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: ml
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ml
  Day 1 (Baseline): number analyzed (Participants) | 29 | 32 | 23
  Day 1 (Baseline) | 66.18 [61.40 to 70.96] | 67.25 [62.49 to 72.02] | 65.09 [59.74 to 70.45]
  Day 28 / Early withdrawal: number analyzed (Participants) | 32 | 28 | 26
  Day 28 / Early withdrawal | 67.97 [63.04 to 72.91] | 71.33 [66.16 to 76.50] | 76.55 [70.52 to 82.57]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 27 | 27 | 18
  Change from baseline (Day 28 / Early withdrawal) | 1.79 [-5.60 to 9.18] | 4.08 [-3.16 to 11.32] | 11.45 [2.73 to 20.18]
  Month 12: number analyzed (Participants) | 28 | 25 | 30
  Month 12 | 74.14 [68.94 to 79.33] | 71.11 [65.62 to 76.60] | 73.12 [67.31 to 78.92]
  Change from baseline (Month 12): number analyzed (Participants) | 24 | 23 | 20
  Change from baseline (Month 12) | 7.95 [0.11 to 15.80] | 3.86 [-3.92 to 11.63] | 8.02 [-0.68 to 16.73]

28. Secondary Outcome: Changes in hsCRP Levels During the Study Compared to Baseline
Description: Change in levels of hsCRP during the study compared to baseline. The reported Least square means and confidence interval were from a repeated measures model on log transformed hsCRP data containing treatment, visit as factors, log transformed baseline hsCRP data as a continuous covariate and treatment by visit as interaction terms.
  For log-transformed data change was defined as division value at corresponding time point and baseline value.
Time Frame: From Day 1 until Day 28
Population: as for outcome 10
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo
Number analyzed (Participants) | 34 | 34 | 33
ratio
  Change from baseline (Day 3) | 2.54 [1.64 to 3.94] | 2.81 [1.81 to 4.35] | 3.75 [2.40 to 5.85]
  Change from baseline (Day 14): number analyzed (Participants) | 31 | 31 | 32
  Change from baseline (Day 14) | 0.31 [0.18 to 0.51] | 0.22 [0.13 to 0.37] | 1.54 [0.92 to 2.59]
  Change from baseline (Day 28 / Early withdrawal): number analyzed (Participants) | 31 | 32 | 32
  Change from baseline (Day 28 / Early withdrawal) | 0.34 [0.20 to 0.58] | 0.23 [0.13 to 0.39] | 0.56 [0.33 to 0.97]

ADVERSE EVENTS:
Time Frame: Information on all Adverse Events (AEs) was collected since signing informed consent form (ICF) and until the study completion by the subject (up to day 365). SAEs for every participant were recorded since his/her signing ICF and for up to 30 days after the study product treatment discontinuation or until the last visit of the participant whichever is the latter, assessed up to 365 days. (AEs recorded prior to the study product administration were added to eCRF section "Medical history".)
Description: Safety set included all randomized subjects, who received the study products (RPH-104 or placebo). This population was used for the safety analysis.
  The tables below show:
  * Treatment-emergent adverse events (TEAEs) - AEs that started at or after the time of application of randomized treatment;
  * Pre-treatment adverse events - AEs that started between the date of signing the ICF by the patient and the time of application of randomized treatment (before receiving any of target treatments).
Groups:
- Pre-treatment Monitoring of "RPH-104 80 mg" Group: subjects randomized to group "RPH-104 80 mg" assessed between the date of the patient being enrolled in the study (by signing the ICF) and the time of application of randomized treatment (before receiving the target treatment)
- Pre-treatment Monitoring of "RPH-104 160 mg" Group: subjects randomized to group "RPH-104 160 mg" assessed between the date of the patient being enrolled in the study (by signing the ICF) and the time of application of randomized treatment (before receiving the target treatment)
- Pre-treatment Monitoring of Placebo Group: subjects randomized to placebo group assessed between the date of the patient being enrolled in the study (by signing the ICF) and the time of application of randomized treatment (before receiving the target treatment)
Arm/Group | RPH-104 80 mg | RPH-104 160 mg | Placebo | Pre-treatment Monitoring of "RPH-104 80 mg" Group | Pre-treatment Monitoring of "RPH-104 160 mg" Group | Pre-treatment Monitoring of Placebo Group
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/34 | 1/34 | 0/34 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 7/34 | 1/34 | 4/34 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 21/34 | 20/34 | 14/34 | 3/34 | 3/34 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPH-104 80 mg (N=34) | RPH-104 160 mg (N=34) | Placebo (N=34) | Pre-treatment Monitoring of "RPH-104 80 mg" Group (N=34) | Pre-treatment Monitoring of "RPH-104 160 mg" Group (N=34) | Pre-treatment Monitoring of Placebo Group (N=34)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPH-104 80 mg (N=34) | RPH-104 160 mg (N=34) | Placebo (N=34) | Pre-treatment Monitoring of "RPH-104 80 mg" Group (N=34) | Pre-treatment Monitoring of "RPH-104 160 mg" Group (N=34) | Pre-treatment Monitoring of Placebo Group (N=34)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (7) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic arteriosclerosis (Vascular disorders) | 6 (6) | 6 (6) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT04463251/Prot_SAP_000.pdf